CLINICAL TRIAL: NCT00331981
Title: Study of the Efficacy and Safety After Long-Term Treatment With Amisulpride in Schizophrenic Patients
Brief Title: Amisulpride in Schizophrenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8968
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Amisulpride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Amisulpride

SUMMARY:
Primary purpose:

* To find out how effective is long term treatment with amisulpride on the positive and negative symptoms in schizophrenic patients
* To find out how safe is long term treatment with amisulpride in schizophrenic patients

Secondary purpose:

* To find out how effective is long term treatment with amisulpride on the quality of life in schizophrenic patients
* To find out how effective is long term treatment with amisulpride on the cognitive function in schizophrenic patients

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as schizophrenia or schizophrenic disorder according to DSM-IV
* Patients who need new anti-psychotic drugs or need to change the medication due to aggravations of symptoms or recurrence

Exclusion Criteria:

* Patients with positive symptoms in whom the disorder does not correspond to schizophrenic criteria. (e.g, schizoaffective disorder)
* Patients hypersensitive to the active ingredient or to other ingredients of the study drug
* Prolactin-dependant tumors, pituitary gland prolactinomas and breast cancer
* Pheochromocytoma or Parkinson's disease
* Pregnancy or breast feeding
* Current or recently withdrawn from drug abuse or alcoholism
* Chronic renal failure and other internal or surgical disease which physician decides will be worsened by trial medication or that will affect the metabolism or effects of the trial medication
* Patients with previous histories and clinical improvement was not seen in spite of treatment with 2 anti-psychotics for over 8 weeks
* Slow heart rate of <55bpm, low blood potassium level, congenital prolongation of the QT interval
* Current treatment with a drug likely to cause markedly slow heart rate(<55bpm), low blood potassium level, slowing of intercardiac condition or prolongation of the QT interval

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138
Dates: Start 2004-02

PRIMARY OUTCOMES:
PANSS scores | at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Won Sik Lee, MD, PhD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Seoul, South Korea